CLINICAL TRIAL: NCT01749657
Title: Kinematic and Kinetic Effects of Orthotic Devices for Subjects With Stage II Posterior Tibial Tendon Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R15AR061737-01A1 (NIH); 1R15AR061737 (NIH)
Record Dates: First submitted 2012-09-18; First posted 2012-12-17 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Posterior Tibial Tendon Dysfunction
Keywords: biomechanics; outcomes; foot; orthotic device
MeSH Terms: conditions — Posterior Tibial Tendon Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Off-the-shelf Device and shoe (Active Comparator): subjects will wear an off-the-shelf orthotic device (AirLift PTTD Brace) and standard Edge shoe (Aetrex Co) for 12 weeks
  Interventions: Device: Arizona
- Custom Device - standard and Shoe (Experimental): subjects will wear a custom (standard) orthotic device (Arizona Co) and Edge shoes (Aetrex Co.) for 12 weeks.
  Interventions: Device: Arizona
- Custom Articulated device and Shoe (Experimental): subjects will wear a custom articulated device (Arizona Co) and Edge shoe (Aetrex Co)for 12 weeks
  Interventions: Device: Arizona
- Custom Extended Device and Shoe (Experimental): subjects will wear a custom extended foot plate orthotic device (Arizona Co) and Edge shoe (Aetrex Co) for 12 weeks.
  Interventions: Device: Arizona

INTERVENTIONS:
Device: Arizona — Compare custom versus off-the-shelf devices for pain and function in subjects with stage II Posterior Tibial Tendon Dysfunction (PTTD).
  Other Names: Arizona Brace (3 different designs) versus AirLift PTTD Brace (DJ Orthopedics - AirCast Co)

SUMMARY:
The lack of high quality evidence to guide conservative care for patients with posterior tibial tendon dysfunction (PTTD) has led to controversy over clinical care. Numerous orthotic devices are available to avoid a costly and debilitating surgery but no consensus on which to use has been made. The current study aims to link biomechanical testing of selected devices to clinical outcomes in subjects with PTTD after wearing a device for 12 weeks.

DETAILED DESCRIPTION:
Orthotic devices serve as essential elements of conservative care programs for posterior tibial tendon dysfunction (PTTD). Data on currently used devices remain limited. Current device designs are restrictive and focus on correction of flatfoot kinematics in subjects with stage II PTTD. Restrictive designs that limit ankle motion may lead to weakness and altered gait dynamics. It remains unclear if less restrictive device designs would be more optimal for subjects with stage II PTTD. The aims of the current proposal are to examine the in-vivo biomechanics of different device designs and to use outcomes to identify the device and design optimal for subjects with stage II PTTD. Research Design: This study will use a laboratory based repeated measures design to explore the function of four different orthotic devices in a sample of 60 subjects with stage II PTTD at baseline. Then each subject will be followed prospectively for 12 weeks while wearing one of the orthotic devices. Clinical outcomes including strength, tendon morphology, and self-reported outcomes will be measured at 12 weeks. Baseline foot kinematics will be collected using a three segment foot model (first metatarsal, calcaneus, tibia) while data on ankle kinetics will be derived from the kinematic data and the ground reaction forces. Impact: There are currently no head-to-head comparisons available among the various devices used in the conservative management of stage II PTTD. The proposed study will provide the necessary controlled data to determine the kinematic and kinetic effects of selected devices and the specific components needed to optimize device design. Outcomes will be used to determine which designs are successful to use clinically.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria Stage II PTTD

  * Swelling
  * Pain with Palpation along the tendon
  * Rearfoot eversion
  * Pain single leg heel raise
  * Flexible flat foot deformity
  * Able to walk 15 m
  * > 40 years of age

Exclusion Criteria:

* Unable to walk 15 m
* Symmes-Weinstein monofilament test 5.06 mm
* Inflammatory arthropathies (e.g. rheumatoid arthritis, psoriasis)
* Co-morbid foot conditions (e.g. hallux rigidis, plantar fasciitis)
* Inability to assume a STN posture

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Foot Function Index - Revised | 12 weeks
  The Foot Function Index - Revised (FFI-R) is a newly published version of the original Foot Function Index (FFI) [45]. The original FFI is a validated, disease specific questionnaire that is widely used to measure foot function and document outcomes in observational studies of PTTD [31, 33]. Rasch analyses for the FFI-R indicated a Pearson reliability of 0.96 and item reliability of 0.93. The domains of the 34 items in the FFI-R questionnaire include pain and stiffness, social/emotional issues, personal disability, and social activity limitation. Although the FFI-R is relatively new, the 23 items from the FFI were the basis for the revised scale. The FFI has been used to measure outcomes for a variety of foot and ankle problems including plantar fasciitis, diabetes, and PTTD [32]. The overall score of the FFI-R will be used as a primary outcome variable while the subscales will be used as secondary outcome variables.

SECONDARY OUTCOMES:
Foot and Ankle Ability Measure | 12 weeks
  Assess the self-reported functional outcomes of patients with primarily foot and ankle pain.
Ankle Strength | 12 weeks
  Compare strength changes over the 12 week intervention. Strength measures will include isometric and isokinetic testing using a Biodex System 3 strength testing system
Hip Strength | 12 weeks
  Compare strength changes over the 12 week intervention. Strength measures will include isometric and isokinetic testing using a Biodex System 3 strength testing system
Deep Posterior Compartment Strength | 12 weeks
  Compare deep posterior compartment strength after 12 weeks across the 4 groups in the study

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Neville, PhD, Principal Investigator — Upstate Medical University
Locations (1):
- Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Background] Neville C, Lemley FR. Effect of ankle-foot orthotic devices on foot kinematics in Stage II posterior tibial tendon dysfunction. Foot Ankle Int. 2012 May;33(5):406-14. doi: 10.3113/FAI.2012.0406. PMID 22735283